CLINICAL TRIAL: NCT01663714
Title: Phase II Multicenter Study of Cyclophosphamide, Vincristine, and Prednisone (CVP) Followed by Iodine-131 Anti-B1 Antibody for Patients With Untreated Low-grade Non-Hodgkin's Lymphoma (NHL).
Brief Title: Open Label Multicenter Study of CVP Followed by Iodine-131 Anti-B1 Antibody for Subjects With Untreated Low-Grade Non Hodgkin's Lymphoma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104514
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Results first posted 2013-04-25 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Non-Hodgkin's Lymphoma; tositumomab and iodine I 131 tositumomab; Bexxar; cycolophosphamide, vacristine, and pednisone
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — COP protocol 2; tositumomab I-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open-label, single arm (Experimental): cycolophosphamide, vacristine, and pednisone (CVP) x6 cycles followed by tositumomab and iodine I 131 tositumomab. CVP will be repeated every 21 days for a total of six cycles. tositumomab and iodine I 131 tositumomab will begin within 56 days following the first day of the sixth cycle of CVP. Patient will undergo two dosing phase for the tositumomab and iodine I 131 tositumomab therapy.
  Interventions: Biological: cycolophosphamide, vacristine, and pednisone (CVP) x6 cycles followed by tositumomab and iodine I 131 tositumomab.

INTERVENTIONS:
Biological: cycolophosphamide, vacristine, and pednisone (CVP) x6 cycles followed by tositumomab and iodine I 131 tositumomab. — cycolophosphamide, vacristine, and pednisone (CVP) x6 cycles followed by tositumomab and iodine I 131 tositumomab. CVP will be repeated every 21 days for a total of six cycles. tositumomab and iodine I 131 tositumomab will begin within 56 days following the first day of the sixth cycle of CVP. Patient will undergo two dosing phase for the tositumomab and iodine I 131 tositumomab therapy.

SUMMARY:
This is a phase II, open-label, multicenter study of the efficacy and safety of sequential administration of CVP x 6 followed by tositumomab and iodine I 131 tositumomab (formerly referred to as tositumomab and iodine I 131 tositumomab). All patients who complete three cycles of CVP, regardless of response, will be eligible for treatment with tositumomab and iodine I 131 tositumomab. Subjects who have rapidly progressive disease prior to completing three cycles of CVP may be removed from study.

In order to proceed to tositumomab and iodine I 131 tositumomab therapy, patients must have completed six cycles of CVP within 20 weeks as described. Patients may proceed to Iodine-131 Anti-B1 Antibody if they have progressive disease documented at the response evaluation following 6 cycles of CVP. In addition, patients must still meet the eligibility inclusion exclusion criteria based upon the week 20 assessments, as applicable. Patients must also have an average of ≤25% bone marrow involved by NHL to receive treatment with tositumomab and iodine I 131 tositumomab. The dosimetric dose of tositumomab and iodine I 131 tositumomab must be given within 28 days of the response evaluation following CVP and no later than 56 days from the first day of the sixth cycle of CVP.

DETAILED DESCRIPTION:
This is a phase II, open-label, multicenter study of the efficacy and safety sequential administration of cycolophosphamide, vacristine, and prednisone (CVP) x6 cycles followed by tositumomab and iodine I 131 tositumomab for previously untreated subjects with low-grade Non-Hodgkin's Lymphoma (NHL). CVP will be repeated every 21 days for a total of six cycles. tositumomab and iodine I 131 tositumomab will begin within 56 days following the first day of the sixth cycle of CVP. Subjects will undergo two dosing phase for the tositumomab and iodine I 131 tositumomab therapy. In the first phase, "dosimetric dose", patients will receive an infusion of unlabeled Anti-B1 Antibody (450mg) over 60 minutes followed by a 30 minute infusion (including a 10-minutes flush) of Anti-B1 (35mg) containing 5mCi of Iodine-131. Whole body gamma camera scans will be obtained on Day 0; Day 2, 3, or 4 and Day 6 or 7 following the dosimetric dose. Using the dosimetric data from three time points, a patient-specific dose of Iodine-131 will be calculated to deliver the desired total body dose of radiotherapy. In the second phase, termed the "therapeutic dose", patients will receive 60-minute infusion of unlabeled Anti-B1 Antibody (450 mg) followed by a 30-minute infusion (including a 10-minute flush) of 35 mg Anti-B1 Antibody labeled with the subjects -specific dose of Iodine-131 calculate to deliver a 75cGy total body radiation dose. Subjects who have platelet counts of 100,000-149,999 cells/mm3 will receive 65 cGy; obese patients will be dosed base upon 137% of their lean body mass. Subjects will be treated with saturated solution potassium iodide (SSKI), Lugol's solution, or potassium iodide tablets starting at least 24 hours prior to the first infusion of the tositumomab and iodine I 131 tositumomab (i.e., the dosimetric dose) and continuing for 14 days following the least infusion of tositumomab and iodine I 131 tositumomab (i.e., the therapeutic dose).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a histologically confirmed initial diagnosis of low-grade non-Hodgkin's B-cell lymphoma according to the International Working Formulation (IWF) (32) (i.e., small lymphocytic with or without plasmacytoid differentiation; follicular small cleaved cell; or follicular, mixed small cleaved and large cell).
* Subjects must have Ann Arbor Stage III, Stage IV, or bulky Stage II disease at diagnosis. Bulky Stage II is defined as a mediastinal mass greater than one-third of the maximum chest diameter, or any other mass greater than or equal to 10 cm in maximum diameter.
* Subjects must have evidence that their tumor tissue expresses the CD20 antigen. Immunoperoxidase stains of paraffin-embedded tissue showing positive reactivity with L26 antibody or immunoperoxidase stains of frozen tissue showing positive reactivity with Anti B1 Antibody (Coulter Clone®) or similar commercially available CD20 antibody or evidence of CD20 positivity by flow cytometry are acceptable evidence of CD20 positivity. Testing of tumor tissue from any time in the course of the patient's disease is acceptable.
* Subjects must have a performance status of at least 60% on the Karnofsky Performance Scale and an anticipated survival of at least 3 months.
* Subjects must have an ANC≥1500 cells/mm3 and a platelet count ≥100,000 cells/mm3 within 14 days of study enrollment. These blood counts must be sustained without support of hematopoietic cytokines or transfusion of blood products.
* Subjects must have adequate renal function (defined as serum creatinine <1.5 times the upper limit of normal) and hepatic function (defined as total bilirubin <1.5 times the upper limit of normal and AST <5 times the upper limit of normal) within 14 days of study enrollment.
* Subjects must have bi-dimensionally measurable disease. At least one lesion must be ≥2.0x2.0 cm by computerized tomography scan.
* Subjects must be at least 18 years of age.
* Subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.
* Subjects must give written informed consent and sign an IRB-approved informed consent form prior to study enrollment.

Exclusion Criteria:

* Subjects who have received prior chemotherapy, biologic therapy, steroids, or radiation therapy as treatment for their NHL.
* Subjects with active obstructive hydronephrosis.
* Subjects with New York Heart Association class III or IV heart disease or other serious illness that would preclude evaluation.
* Subjects with prior malignancy other than lymphoma, except for adequately treated skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years. Patients who have been disease-free of another cancer for greater than 5 years must be carefully assessed at the time of study entry to rule out recurrent disease.
* Subjects with known HIV infection.
* Subjects who are HAMA positive.
* Subjects with known brain or leptomeningeal metastases.
* Subjects who are pregnant or breastfeeding. Males and females must agree to use a contraceptive method from enrollment to 6 months after receiving Iodine 131 Anti B1 Antibody.
* Subjects with active infection requiring IV anti-infectives at the time of study enrollment.
* Subjects with intermediate- or high-grade NHL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Link BK, Martin P, Kaminski MS, Goldsmith SJ, Coleman M, Leonard JP. Cyclophosphamide, vincristine, and prednisone followed by tositumomab and iodine-131-tositumomab in patients with untreated low-grade follicular lymphoma: eight-year follow-up of a multicenter phase II study. J Clin Oncol. 2010 Jun 20;28(18):3035-41. doi: 10.1200/JCO.2009.27.8325. Epub 2010 May 10. PMID 20458031
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 104514 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104514 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104514 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104514 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104514 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104514 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104514 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) received cyclophosphamide (C), vincristine (V), prednisone (P) in the first study phase (P). Upon completion of this P, par. began the first of 2 phases of radio immunotherapy: P1, dosimetric dose (DD); P2, therapeutic dose. Par. completing 2 years of the study could enter a long-term follow-up study (BEX104528; NCT00240578).
Groups:
- Chemotherapy; TST and Iodine I 131 TST: Par. received 6 cycles of chemotherapy (chemo.): oral Cyclophosphamide (400 milligrams/meters squared [mg/m^2]/day) for 1-5 days; intravenous (IV) Vincristine (1.4 mg/m^2) on Day 1; oral Prednisone (100 mg/m^2/day) for 1-5 days. Par. received the DD 4-8 weeks after Day 1 of Cycle 6 of chemo. Unlabeled tositumomab (TST) (450 mg) was infused IV for 1 hour prior to a 30 minute infusion of 35 mg TST trace labeled with 5 millicurie (mCi) Iodine 131. Par. received 4 drops by mouth (DBM) 3 times a day (TID) of potassium iodide (KI) and 20 DBM TID Lugol's solution or KI tablets (130 mg BM, daily) >=24 hours prior to DD administration.Treatment continued daily for 14 days after the therapeutic dose (TD: a 1 hour IV infusion of 450 mg TST), followed by an infusion of 35 mg TST radiolabeled with Iodine I 131 to deliver a 75 centiGray total body radiation dose. Par. completing 2 years of the study could enter a 10-year Long-Term Follow-Up study (BEX104528) in which no study medication was given.
Period: Dosimetric and Therapeutic Treatment
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Started | 30
Completed | 0
Not Completed | 30
Not completed — Lost to Follow-up | 3
Not completed — Progressive Disease | 11
Not completed — Rolled Over to Study BEX104528 | 16
Period: Long-Term Follow-Up
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Started | 22 (22 of the30 participants withdrawing from Study BEX104514 enrolled in the LTFU study.)
Completed | 16
Not Completed | 6
Not completed — Lost to Follow-up | 1
Not completed — Death | 4
Not completed — Non-compliance | 1

BASELINE CHARACTERISTICS:
Groups:
- Chemotherapy; TST and Iodine I 131 TST: Par. received 6 cycles of chemo.: oral Cyclophosphamide (400 mg/m^2/day) for 1-5 days; IV Vincristine (1.4 mg/m^2) on Day 1; oral Prednisone (100 mg/m^2/day) for 1-5 days. Par. received the DD 4-8 weeks after Day 1 of Cycle 6 of chemo. Unlabeled TST (450 mg) was infused IV for 1 hour prior to a 30 minute infusion of 35 mg TST trace labeled with 5 mCi Iodine 131. Par. received 4 DBM TID of KI and 20 DBM TID Lugol's solution or KI tablets (130 mg BM, daily) >=24 hours prior to DD administration.Treatment continued daily for 14 days after the TD: a 1 hour IV infusion of 450 mg TST, followed by an infusion of 35 mg TST radiolabeled with Iodine I 131 to deliver a 75 centiGray total body radiation dose. Par. completing 2 years of the study could enter a 10-year Long-Term Follow-Up study (BEX104528) in which no study medication was given.
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.6 (9.5)
Gender [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Race/Ethnicity, Customized [Number; unit: participants]
  White | 28
  Hispanic | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Par.) With Unconfirmed Response (Complete Response, Complete Response/Unconfirmed, or Partial Response), as Assessed by the Investigator
Description: Par. with response include those with Complete Response (CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease), Complete Response/unconfirmed (CRu: complete resolution of all disease-related symptoms; residual lymph node mass >1.5 centimeters in the greatest transverse diameter that has regressed by >75%, indeterminate bone marrow, are present), or Partial Response (PR: >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions; no new lesions).
Time Frame: Par. were evaluated until death/disease progression or for 2 years in Study BEX104514. Par. who completed 2 years in Study BEX104514 were followed in Study BEX104528 for up to 130 months. Data are included from Study BEX104514 and Study BEX104528.
Population: Intent-to-Treat (ITT) Exposed Population: all participants who were enrolled into the study and received at least one dose of study drug. Only those participants evaluable for response were analyzed.
Measure: Number; unit: participants
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
participants | 30
Statistical Analysis 1: Comparison: Chemotherapy; TST and Iodine I 131 TST; Test type: Superiority or Other; percentage of participants = 100, 95% CI 2-sided [100 to 100] — The estimated value represents the percentage of participants with unconfirmed response

2. Primary Outcome: Number of Participants (Par.) With Confirmed Response (Complete Response [CR], Complete Response/Unconfirmed [CRu], or Partial Response [PR]), as Assessed by the Investigator
Description: CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease. CRu: complete resolution of all disease-related symptoms; residual lymph node mass >1.5 centimeters in the greatest transverse diameter that has regressed by >75%, indeterminate bone marrow, are present. PR: >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions; no new lesions. Confirmed response required CR, CRu, or PR, which were confirmed by 2 separate response evaluations >=4 weeks apart.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
participants | 30
Statistical Analysis 1: Comparison: Chemotherapy; TST and Iodine I 131 TST; Test type: Superiority or Other; percentage of participants = 100, 95% CI 2-sided [100 to 100] — The estimated value represents the percentage of participants with confirmed response

3. Secondary Outcome: Number of Participants With Unconfirmed Complete Response (CR), as Assessed by the Investigator
Description: CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease, if present before therapy.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Number; unit: participants
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
participants | 21

4. Secondary Outcome: Number of Participants With Confirmed Complete Response (CR), as Assessed by the Investigator
Description: CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease, if present before therapy. Confirmed response required CR, which was confirmed by 2 separate response evaluations >=4 weeks apart.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Number; unit: participants
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
participants | 21

5. Secondary Outcome: Duration of Response (DOR), as Assessed by the Investigator
Description: DOR=the time from the first documented response (for par. with CR, CRu, or PR) until disease progression (DP). DP=a >=50% increase from the nadir value (lowest laboratory value recorded following administration of study medication) of the sum of the products of the longest perpendicular diameters of all measurable lesions or the appearance of any new lesion. Individual lesions must be >1.5 centimeters (cm) in diameter by radiographic evaluation or >1 cm in diameter by physical examination. Responses had to be confirmed by 2 separate evaluations occurring >=4 weeks apart.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants with response were analyzed. Participants who did not experience progression were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 14
months
  Unconfirmed Responders | 129.6 [42.1 to NA] — There were not enough events of progression to be able to determine/calculate the upper limit of the 95% confidence interval (CI).
  Confirmed Responders | 129.6 [42.1 to NA] — There were not enough events of progression to be able to determine/calculate the upper limit of the 95% CI.

6. Secondary Outcome: DOR for Unconfirmed and Confirmed Complete Response, as Assessed by the Investigator
Description: DOR=the time from the first documented response (for par. with CR) until disease progression (DP). DP=a >=50% increase from the nadir value (lowest laboratory value recorded following administration of study medication) of the sum of the products of the longest perpendicular diameters of all measurable lesions or the appearance of any new lesion. Individual lesions must be >1.5 centimeters (cm) in diameter by radiographic evaluation or >1 cm in diameter by physical examination. Responses had to be confirmed by 2 separate evaluations occurring >=4 weeks apart.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 7
months
  Unconfirmed Responders with CR | 129.6 [74.8 to NA] — There were not enough events of progression to be able to determine/calculate the upper limit of the 95% CI.
  Confirmed Responders with CR | 129.6 [74.8 to NA] — There were not enough events of progression to be able to determine/calculate the upper limit of the 95% CI.

7. Secondary Outcome: Time to Progression of Disease or Death, as Assessed by the Investigator
Description: Time to progression or progression-free survival is defined as the time from the dosimetric dose to the first documented occurrence of disease progression or death. Disease progression is defined as a >=50% increase from the nadir value (lowest laboratory value recorded following administration of the study medication) of the sum of the products of the longest perpendicular diameters of all measurable lesions or the appearance of any new lesion. Individual lesions must be >1.5 cm in diameter by radiographic evaluation or >1 cm in diameter by physical examination.
Time Frame: as for outcome 1
Population: ITT Exposed Population. If a participant did not have progression or did not die, that participant was censored in the survival analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
months | 110.2 [38.3 to NA] — There were not enough events of progression to be able to determine/calculate the upper limit of the 95% CI.

8. Secondary Outcome: Time to Treatment Failure, as Assessed by the Investigator
Description: Time to treatment failure is defined as the time from the start of treatment to the first occurrence of study withdrawal, progression, or death.
Time Frame: as for outcome 1
Population: ITT Exposed Population. If a participant did not have treatment failure, that participant was censored in the survival analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
months | 78.9 [36.5 to NA] — There were not enough events to be able to determine/calculate the upper limit of the 95% CI.

9. Secondary Outcome: Total Body Residence Time (TBRT; Average Amount of Time TST Spends in the Body, Calculated From the Rate of TB Clearance of Radioactivity During the Dosimetric Dose [DD]) of Iodine 131 TST Antibody Following the DD
Description: To determine TBRT, the percent-injected activity (PIA) is calculated from the background-corrected (BC) total body count (TBC) at D 0; D 2/3/4; and D 7. The time from the DD to the acquisition of whole body count (WBC) is then determined. The PIA remaining at each time point (TP) is then calculated by dividing the BC WBC for that TP by the BC WBC from the first TP (D 0) * 100. To determine RT, a best-fit line from 100% (pre-plotted D 0 value) through 2 plotted points (other TPs) is made. TBRT=the x-axis value at the point where the line intersects the horizontal 37% injected activity line.
Time Frame: Day (D) 0; D 2, 3, or 4; and D 6 or 7
Population: ITT Exposed Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
hours | 103.7 (8.55)

10. Secondary Outcome: Time to Nadir for Hematological Parameters: Absolute Neutrophil Count (ANC), Hemoglobin, Platelets, and White Blood Cell (WBC) Count
Description: Nadir is defined as the lowest laboratory value recorded up to 120 days following the therapeutic dose (or the dosimetric dose for participants who did not receive the therapeutic dose).
Time Frame: Up to 120 days following the therapeutic dose (given on Study Day 7, following the dosimetric dose) (or the dosimetric dose for participants who did not receive the therapeutic dose)
Population: ITT Exposed Population
Measure: Median (Full Range); unit: days
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
days
  ANC | 49.0 [15 to 78]
  Hemoglobin | 49.0 [34 to 85]
  Platelets | 35.5 [26 to 56]
  WBC count | 44.0 [15 to 78]

11. Secondary Outcome: Time to Recovery (TTR) to Baseline (BL) for Hematologic Laboratory (Lab.) Evaluations
Description: TTR to BL grade (gr.) for par. with a Gr. 0 toxicity (tox.=lab. value outside the normal range) at BL=time from the last administration of study drug (SD) to the first post-nadir (PN) date with Gr. 0 toxicity with no other Gr. 1-4 toxicities recorded within the next week. For par. with a higher gr. tox. at BL, TTR=time from the last administration of SD to the first PN date with the BL gr. or better with no other higher gr. toxicities recorded during the next week. Each lab. established its own reference range using data from its own equipment/methods; there is no standard reference range.
Time Frame: as for outcome 10
Population: ITT Exposed Population. Only those participants with hematologic toxicity were evaluated for time to recovery to baseline.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
days
  Time to recovery to baseline ANC, n=30 | 77.0 [70.0 to 91.0]
  Time to recovery to baseline hemoglobin, n=28 | 76.5 [62.0 to 168.0]
  Time to recovery to baseline platelets, n=30 | 60.5 [50.0 to 75.0]
  Time to recovery to baseline WBC count, n=29 | 126.5 [75.0 to 170.0]

12. Secondary Outcome: Nadir Values for Absolute Neutrophil Count (ANC)
Description: as for outcome 10
Time Frame: as for outcome 10
Population: ITT Exposed Population
Measure: Median (Full Range); unit: 10^3 cells/cubic millimeters (mm^3)
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
10^3 cells/cubic millimeters (mm^3) | 0.4 [0 to 4]

13. Secondary Outcome: Nadir Values for Hemoglobin
Description: as for outcome 10
Time Frame: as for outcome 10
Population: ITT Exposed Population
Measure: Median (Full Range); unit: Grams/deciliter (g/dL)
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
Grams/deciliter (g/dL) | 10.6 [6 to 15]

14. Secondary Outcome: Nadir Values for Platelet Count
Description: as for outcome 10
Time Frame: as for outcome 10
Population: ITT Exposed Population
Measure: Median (Full Range); unit: 10^3 cells/microliter (µL)
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
10^3 cells/microliter (µL) | 57.0 [4 to 145]

15. Secondary Outcome: Nadir Values for WBC Count
Description: as for outcome 10
Time Frame: as for outcome 10
Population: ITT Exposed Population
Measure: Median (Full Range); unit: 10^3 cells/µL
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
10^3 cells/µL | 1.8 [0 to 5]

16. Secondary Outcome: Number of Participants With the Indicated Grade 3 or Grade 4 Adverse Events (AEs)
Description: AEs were graded using the Common Toxicity Criteria from the Cancer Therapy Evaluation Program, Division of Cancer Therapy, National Cancer Institute. Grades: 0 = No AE or within normal limits; 1 = Mild AE; 2 = Moderate AE; 3 = Severe and undesirable AE; 4 = Life-threatening or disabling AE; 5 = Death related to AE.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Number; unit: participants
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
participants
  ANC <1000 cells/mm^3 | 29
  WBC <2000 cells/mm^3 | 23
  Platelets <50000 cells/mm^3 | 12
  Hemoglobin <8.0 g/dL | 2
  Neutropenia | 15
  Leukopenia | 6
  Febrile neutropenia | 5
  Thrombocytopenia | 4
  Anemia | 3
  Granulocytopenia | 1
  Lymphopenia | 1
  Alopecia | 9
  Night sweats | 1
  Acute myeloid leukaemia | 2
  Basal cell carcinoma | 2
  Myelodysplastic syndrome | 1
  Prostate cancer | 1
  Squamous cell carcinoma | 1
  Perirectal abscess | 2
  Urinary tract infection | 2
  Cystitis | 1
  Neutropenic infection | 1
  Otitis media | 1
  Periorbital cellulitis | 1
  Aphasia | 1
  Cerebrovascular accident | 1
  Headache | 1
  Hypoaesthesia | 1
  VIIth nerve paralysis | 1
  Asthenia | 1
  Pyrexia | 1
  Myalgia | 1
  Pain in extremity | 1
  Depression | 1
  Insomnia | 1
  Amenorrhoea | 1
  Breast mass | 1
  Conjunctivitis | 1
  Constipation | 1
  Drug hypersensitivity | 1
  Aspartate aminotransferase increased | 1
  Cystitis hemorrhagic | 1
  Epistaxis | 1

17. Secondary Outcome: Number of Participants With the Indicated Grade 3 or Grade 4 AEs Possibly or Probably Related to Study Drug
Description: AEs were graded using the Common Toxicity Criteria from the Cancer Therapy Evaluation Program, Division of Cancer Therapy, National Cancer Institute. Grades: 0 = No AE or within normal limits; 1 = Mild AE; 2 = Moderate AE; 3 = Severe and undesirable AE; 4 = Life-threatening or disabling AE; 5 = Death related to AE. The Investigator assessed whether the AE was possibly or probably related to study drug. In addition, all laboratory-derived hematologic toxicities (values outside the normal range) were assumed to be possibly or probably related to study drug.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Number; unit: participants
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
participants
  ANC <1000 cells/mm^3 | 29
  WBC <2000 cells/mm^3 | 23
  Platelets <50000 cells/mm^3 | 12
  Hemoglobin <8.0 g/dL | 2
  Neutropenia | 15
  Leukopenia | 6
  Febrile neutropenia | 5
  Thrombocytopenia | 4
  Anemia | 3
  Granulocytopenia | 1
  Lymphopenia | 1
  Alopecia | 9
  Night sweats | 1
  Perirectal abscess | 2
  Urinary tract infection | 2
  Cystitis | 1
  Neutropenic infection | 1
  Otitis media | 1
  Periorbital cellulitis | 1
  Acute myeloid leukaemia | 2
  Basal cell carcinoma | 1
  Myelodysplastic syndrome | 1
  Squamous cell carcinoma | 1
  Headache | 1
  VIIth nerve paralysis | 1
  Depression | 1
  Insomnia | 1
  Conjunctivitis | 1
  Constipation | 1
  Pyrexia | 1
  Aspartate aminotransferase increased | 1
  Myalgia | 1
  Cystitis hemorrhagic | 1
  Amenorrhoea | 1
  Epistaxis | 1

18. Secondary Outcome: Number of Participants With Any Treatment-related Serious Adverse Event (SAE)
Description: An SAE is defined as any event occurring at any dose that results in any of the following outcomes: death, a life-threatening adverse drug experience (at immediate risk of death from the experience as it occurred), inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life threatening, or require hospitalization may be considered to be a serious adverse drug experience when based upon appropriate medical judgment.
Time Frame: as for outcome 1
Population: ITT-Exposed Population. All participants who experienced a treatment-related SAE were analyzed.
Measure: Number; unit: participants
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 11
participants
  Febrile neutropenia | 5
  Anaemia | 2
  Neutropenia | 2
  Thrombocytopenia | 2
  Granulocytopenia | 1
  Leukopenia | 1
  Acute myeloid leukaemia | 2
  Basal cell carcinoma | 1
  Myelodysplastic syndrome | 1
  Squamous cell carcinoma | 1
  Perirectal abscess | 2
  Neutropenic infection | 1
  Pyrexia | 1
  Cystitis hemorrhagic | 1

19. Secondary Outcome: Number of Participants With the Indicated Primary Cause of Death
Description: The primary cause of death of the participants was assessed by the Investigator.
Time Frame: as for outcome 1
Population: ITT Exposed Population. All participants who died during the study were analyzed.
Measure: Number; unit: participants
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 9
participants
  Progression of lymphoma | 5
  Complications related to study drug | 1
  Other | 3

20. Secondary Outcome: Number of Participants Who Received Any Supportive Care
Description: Supportive care is defined as interventions that help the participants achieve comfort but do not affect the course of a disease.
Time Frame: as for outcome 1
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
participants | 17

21. Secondary Outcome: Number of Participants Who Were Negative for Human Anti-murine Antibodies (HAMA) at Baseline (Study Entry) But Positive or Negative at Month 24
Description: The administration of murine antibodies may form HAMA. A HAMA assay was performed using the ImmunoSTRIP HAMA IgG enzyme-linked immune absorbent assay by a central laboratory (Covance Classic Laboratory Services, Indianapolis, IN). To be "positive," a participant had to have a positive HAMA assessment during the first 24 months.
Time Frame: Day 1 to Day 730 (24 months) after receiving the dosimetric dose
Population: ITT Exposed Population
Measure: Number; unit: participants
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 30
participants
  Positive | 0
  Negative | 30

22. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the treatment start date to the date of death from any cause.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy; TST and Iodine I 131 TST
Number analyzed (Participants) | 9
months | NA [NA to NA] — There were not enough events to be able to calculate the median or the confidence interval.

ADVERSE EVENTS:
Time Frame: Par. were evaluated until death/disease progression or for 2 years in Study BEX104514. Par. who completed 2 years in Study BEX104514 were followed in Study BEX104528 for up to 130 months. Data are included from both Study BEX104514 and Study BEX104528.
Groups:
- Period After CVP: Par. received 6 cycles of chemotherapy as follows: oral Cyclophosphamide (400 mg/m^2/day) for 1-5 days; intravenous Vincristine (1.4 mg/m^2) on Day 1; oral Prednisone (100 mg/m^2/day) for 1-5 days
- Period After Dosimetric and Therapeutic Dose: After receiving Cyclophosphamide, Vincristine, and Prednisone, par. received the DD 4-8 weeks after Day 1 of Cycle 6 of chemo. Unlabeled tositumomab (TST) (450 mg) was infused IV for 1 hour prior to a 30 minute infusion of 35 mg TST trace labeled with 5 millicurie (mCi) Iodine 131. Par. received 4 drops by mouth (DBM) 3 times a day (TID) of potassium iodide (KI) and 20 DBM TID Lugol's solution or KI tablets (130 mg BM, daily) >=24 hours prior to DD administration.Treatment continued daily for 14 days after the therapeutic dose (TD: a 1 hour IV infusion of 450 mg TST), followed by an infusion of 35 mg TST radiolabeled with Iodine I 131 to deliver a 75 centiGray total body radiation dose.
- Combined Regimen Period: Par. received 6 cycles of chemo.: oral Cyclophosphamide (400 mg/m^2/day) for 1-5 days; IV Vincristine (1.4 mg/m^2) on Day 1; oral Prednisone (100 mg/m^2/day) for 1-5 days. Par. received the DD 4-8 weeks after Day 1 of Cycle 6 of chemo. Unlabeled TST (450 mg) was infused IV for 1 hour prior to a 30 minute infusion of 35 mg TST trace labeled with 5 mCi Iodine 131. Par. received 4 DBM TID of KI and 20 DBM TID Lugol's solution or KI tablets (130 mg BM, daily) >=24 hours prior to DD administration.Treatment continued daily for 14 days after the TD: a 1 hour IV infusion of 450 mg TST, followed by an infusion of 35 mg TST radiolabeled with Iodine I 131 to deliver a 75 centiGray total body radiation dose. Par. completing 2 years of the study could enter a 10-year Long-Term Follow-Up study (BEX104528) in which no study medication was given.
Arm/Group | Period After CVP | Period After Dosimetric and Therapeutic Dose | Combined Regimen Period
Serious Adverse Events (participants affected / at risk) | 7/30 | 8/30 | 13/30
Other Adverse Events (participants affected / at risk) | 30/30 | 30/30 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period After CVP (N=30) | Period After Dosimetric and Therapeutic Dose (N=30) | Combined Regimen Period (N=30)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 0 | 5
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 2
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Perirectal abscess (Infections and infestations) | 2 | 0 | 2
Neutropenic infection (Infections and infestations) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Cystitis hemorrhagic (Renal and urinary disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period After CVP (N=30) | Period After Dosimetric and Therapeutic Dose (N=30) | Combined Regimen Period (N=30)
ANC <1000 cells/mm^3 (Investigations) | 25 | 15 | 29
WBC <2000 cells/mm^3 (Investigations) | 16 | 17 | 23
Platelets <50000 cells/mm^3 (Investigations) | 1 | 12 | 12
Hemoglobin <8.0 g/dL (Investigations) | 0 | 2 | 2
Fatigue (General disorders) | 14 | 15 | 23
Pyrexia (General disorders) | 6 | 2 | 7
Chills (General disorders) | 3 | 4 | 7
Asthenia (General disorders) | 6 | 0 | 6
Pain (General disorders) | 3 | 1 | 4
Edema peripheral (General disorders) | 2 | 1 | 3
Chest discomfort (General disorders) | 0 | 1 | 1
Chest pain (General disorders) | 0 | 1 | 1
Crepitations (General disorders) | 1 | 0 | 1
Facial pain (General disorders) | 1 | 0 | 1
Feeling hot (General disorders) | 1 | 0 | 1
Ill-defined disorder (General disorders) | 0 | 1 | 1
Malaise (General disorders) | 1 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 1
Nodule (General disorders) | 1 | 0 | 1
Suprapubic pain (General disorders) | 1 | 0 | 1
Xerosis (General disorders) | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 21 | 1 | 21
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 1 | 5
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Swelling face (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin tightness (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 13 | 13
Headache (Nervous system disorders) | 7 | 3 | 10
Paraesthesia (Nervous system disorders) | 5 | 2 | 7
Dizziness (Nervous system disorders) | 2 | 1 | 3
Dysgeusia (Nervous system disorders) | 3 | 0 | 3
Hypoaesthesia (Nervous system disorders) | 3 | 0 | 3
Neuropathy peripheral (Nervous system disorders) | 3 | 0 | 3
Aphasia (Nervous system disorders) | 1 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 1
Hyporeflexia (Nervous system disorders) | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1
Sinus headache (Nervous system disorders) | 1 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 15 | 3 | 16
Diarrhea (Gastrointestinal disorders) | 6 | 2 | 8
Constipation (Gastrointestinal disorders) | 7 | 0 | 7
Stomatitis (Gastrointestinal disorders) | 6 | 0 | 6
Abdominal distension (Gastrointestinal disorders) | 4 | 1 | 5
Abdominal discomfort (Gastrointestinal disorders) | 3 | 2 | 4
Vomiting (Gastrointestinal disorders) | 3 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 2 | 2
Oral pain (Gastrointestinal disorders) | 2 | 0 | 2
Tooth disorder (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 1
Anal pruritus (Gastrointestinal disorders) | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 1
Oral disorder (Gastrointestinal disorders) | 0 | 1 | 1
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Salivary gland disorder (Gastrointestinal disorders) | 1 | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 1 | 0 | 1
Tongue discolouration (Gastrointestinal disorders) | 1 | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 21 | 3 | 21
Leukopenia (Blood and lymphatic system disorders) | 8 | 3 | 8
Anaemia (Blood and lymphatic system disorders) | 6 | 1 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0 | 2
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 6
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal mucosal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 3 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 3 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 0 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle hypertrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 2 | 5
Nasopharyngitis (Infections and infestations) | 2 | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 3
Bronchitis (Infections and infestations) | 1 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 1
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 6 | 1 | 7
Anxiety (Psychiatric disorders) | 3 | 1 | 4
Depression (Psychiatric disorders) | 3 | 0 | 3
Restlessness (Psychiatric disorders) | 1 | 1 | 2
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 1
Emotional distress (Psychiatric disorders) | 1 | 0 | 1
Hypervigilance (Psychiatric disorders) | 1 | 0 | 1
Mood altered (Psychiatric disorders) | 1 | 0 | 1
Mood swings (Psychiatric disorders) | 1 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 1 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 4 | 2 | 6
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 1
Bladder irritation (Renal and urinary disorders) | 1 | 0 | 1
Bladder pain (Renal and urinary disorders) | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0 | 1
Blood bicarbonate decreased (Investigations) | 2 | 0 | 2
Weight decreased (Investigations) | 1 | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Blood potassium increased (Investigations) | 1 | 0 | 1
Blood sodium decreased (Investigations) | 1 | 0 | 1
Body temperature decreased (Investigations) | 1 | 0 | 1
Body temperature increased (Investigations) | 0 | 1 | 1
Cardiac murmur (Investigations) | 0 | 1 | 1
Heart rate increased (Investigations) | 1 | 0 | 1
Heart rate irregular (Investigations) | 0 | 1 | 1
Weight increased (Investigations) | 1 | 0 | 1
Amenorrhea (Reproductive system and breast disorders) | 3 | 0 | 3
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 1
Vision blurred (Eye disorders) | 2 | 0 | 2
Conjunctivitis (Eye disorders) | 1 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 1
Keratitis (Eye disorders) | 1 | 0 | 1
Varicose vein (Vascular disorders) | 1 | 1 | 2
Flushing (Vascular disorders) | 1 | 0 | 1
Hematoma (Vascular disorders) | 0 | 1 | 1
Phlebitis (Vascular disorders) | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 1
Hypogammaglobulinaemia (Immune system disorders) | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 1
Cushingoid (Endocrine disorders) | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.